CLINICAL TRIAL: NCT04474665
Title: A Single-arm, Prospective Study of Tornier Blueprint Planning Software in Patients Receiving Reverse Shoulder Arthroplasty
Brief Title: Tornier Blueprint Planning Software in Patients Receiving Reverse Shoulder Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Spine Institute of Louisiana Foundation (Industry)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Blueprint-2019
Record Dates: First submitted 2020-07-08; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Reverse Shoulder Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Implant placement accuracy (Other): Blueprint planning software will be used to plan reverse shoulder replacement surgery. Accuracy of the placement compared to the plan will be assessed post-surgery.
  Interventions: Device: Reverse shoulder arthroplasty utilizing Blueprint Software

INTERVENTIONS:
Device: Reverse shoulder arthroplasty utilizing Blueprint Software — Reverse shoulder arthroplasty utilizing Blueprint Software

SUMMARY:
Compare sizing determined in pre-operative planning of reverse shoulder arthroplasty to operative implant size selected.

DETAILED DESCRIPTION:
The Blueprint planning software automatically creates a virtual implantation environment for the surgeon to use. The use of 3D measurements is independent of patient positioning, which results in more accurate measurements of the glenoid version and inclination measurements in shoulder replacement surgery.

Pre-operative planning with Blueprint can accurately predict intraoperative implant selection within one size. Also, pre-operative planning leads to case efficiency and improved functional outcomes at 6 months post-operative compared to Baseline.

The objective of this study is to characterize implant size accuracy, planning time, functional outcomes, and procedural time (i.e., surgical time) using Blueprint planning software in subjects who are candidates for reverse shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature, and age ≥ 18 years.
2. In the opinion of the treating surgeon, must already be a qualified candidate for reverse shoulder arthroplasty without the use of glenoid bone grafts.
3. Be likely to return for regular follow-ups until the end of the study period.
4. Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria:

1. Previous bony surgery on the operative shoulder.
2. Shoulder pain due to acute trauma.
3. Clinical, laboratory and/or radiological evidence of shoulder pain secondary to acute or chronic infection, malignancy, other space occupying lesions and metabolic bone demineralization diseases (e.g. osteomalacia, gout, Paget's disease etc.)
4. Any active malignancy, infectious process, or documented chronic autoimmune disease.
5. Any other concurrent medical disease or treatment that might impair normal healing process.
6. Recent history (within past 6 months) of any chemical or alcohol dependence.
7. Currently a prisoner.
8. Currently experiencing a major mental illness (psychosis, schizophrenia, major affective disorder) which may indicate that the symptoms are psychological rather than of physical origin.
9. Pregnant or planning to become pregnant within study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Range of motion | 6 months
  Range of motion of the operative shoulder
Accuracy of sizing | Perioperative
  Blueprint planned implant size compared to actual implant size
Time to plan/perform case | Pre-operative
  Time required for surgeon to plan and perform the case using the Bluerpint software
Time to plan/perform case | Perioperative
  Time required for surgeon to plan and perform the case using the Bluerpint software

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | 12 weeks
  Questionnaire to score and understand how well you function in everyday life, concerning your shoulder pain/limitations. 0-100 score, with higher score indicating higher functionality.
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES) | 6 months
  Questionnaire to score and understand how well you function in everyday life, concerning your shoulder pain/limitations. 0-100 score, with higher score indicating higher functionality.
Simple Shoulder Test (SST) Questionnaire | Pre-operative
  12 yes/no questions to understand your daily functionality concerning your shoulder.
Simple Shoulder Test (SST) Questionnaire | 2 weeks
  12 yes/no questions to understand your daily functionality concerning your shoulder.
Simple Shoulder Test (SST) Questionnaire | 6 weeks
  12 yes/no questions to understand your daily functionality concerning your shoulder.
Simple Shoulder Test (SST) Questionnaire | 12 weeks
  12 yes/no questions to understand your daily functionality concerning your shoulder.
Simple Shoulder Test (SST) Questionnaire | 6 months
  12 yes/no questions to understand your daily functionality concerning your shoulder.
Patient Satisfaction | 12 weeks
  Patient rated satisfaction with surgical treatment rated; very satisfied, somewhat satisfied, somewhat dissatisfied, or very dissatisfied
Patient Satisfaction | 6 months
  Patient rated satisfaction with surgical treatment rated; very satisfied, somewhat satisfied, somewhat dissatisfied, or very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: David Googe, MD, Principal Investigator — Orthopedics Specialists of Louisiana
Locations (1):
- Spine Institute of Louisiana, Shreveport, Louisiana, United States